CLINICAL TRIAL: NCT03821701
Title: A Multicenter, Randomized Controlled Trial of Angiotensin-Neprilysin Inhibition (ARNI) in the Chronic Heart Failure
Brief Title: Effect of Angiotensin-Neprilysin Inhibition (ARNI) on Prognosis of Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Baoji Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2018-019
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Chronic Heart Failure
Keywords: Shakurba valsartan; Heart failure; ACEI/ARB
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Newly diagnosed HFrEF ARNI (Experimental): Newly diagnosed HFrEF patients will be administered ARNI Entresto according to the clinical condition among the whole study.
  Interventions: Drug: Entresto
- Newly diagnosed HFrEF ACEI/ARB (Active Comparator): Newly diagnosed HFrEF patients will be administered ACEI/ARB according to the clinical condition among the whole study.
  Interventions: Drug: ACEI/ARB
- Prior diagnosed HFrEF ARNI (Experimental): Prior diagnosed HFrEF patients will be administered ARNI Entresto according to the clinical condition among the whole study.
  Interventions: Drug: Entresto
- Prior diagnosed HFrEF ACEI/ARB (Active Comparator): Prior diagnosed HFrEF patients will be administered ACEI/ARB according to the clinical condition among the whole study.
  Interventions: Drug: ACEI/ARB

INTERVENTIONS:
Drug: Entresto — Sacubitril Valsartan Sodium Tablets, 100mg bid, among whole study
  Arms: Newly diagnosed HFrEF ARNI; Prior diagnosed HFrEF ARNI
Drug: ACEI/ARB — Choose one of ACEI/ARB according to the clinical condition among the whole study.
  Arms: Newly diagnosed HFrEF ACEI/ARB; Prior diagnosed HFrEF ACEI/ARB

SUMMARY:
This study is a randomized controlled multicenter clinical trial, in which about 340 patients with newly diagnosed or prior diagnosed chronic heart will be recruited. Patients will be randomly divided into Angiotensin-Neprilysin Inhibition (ARNI) group and angiotensin-converting enzyme inhibitors or angiotensin receptor blockers (ACEI/ARB) group. All-cause death, cardiac death and re-hospitalization due to heart failure will be evaluated in 1, 3, 6, 12 months after recruitment.

DETAILED DESCRIPTION:
Chronic heart failure is associated with poor prognosis in cardiac patients, although systemic effective drugs has been applied in these patients. European Society of Cardiology (ESC) has recommended ARNI Sacubitril/Valsartan as first-line drugs in replacement of ACEI (I, B) in 2016 for these patients. While American College of Cardiology and The American Heart Association (ACC/AHA) made a first-line recommendation that patients with heart failure due to reduced ejection fraction (HFrEF) could be administrated ARNI directly. Hence, we apply this trial to find if ARNI could replace ACEI/ARB to provide insights for better treatment of chronic heart failure in China. This study is a randomized controlled multicenter clinical trial, in which about 340 patients with newly diagnosed or prior diagnosed chronic heart will be recruited. Patients will be randomly divided into Angiotensin-Neprilysin Inhibition (ARNI) group and ACEI/ARB group. All-cause death, cardiac death and re-hospitalization due to heart failure will be evaluated in 1, 3, 6, 12 months after recruitment. Other safety assessment including left ventricular ejection fraction (LVEF), 6 minutes walk test will be followed up as well.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* HFrEF, defined as LVEF≤40% and New York Heart Association (NYHA) class ≥ II.
* Plasma NT-proBNP ≥ 600 pg/ml, or NT-proBNP ≥ 400 pg/ml if patients have been hospitalized for heart failure in 12 months.
* If patients have been taking ACEI/ARB at recruitment, a stable dose equivalent to at least 10mg/day of enalapril will be required.
* Volunteer for the study and sign the informed consent.

Exclusion Criteria:

* Symptomatic hypotension, systolic blood pressure < 95 mmHg at baseline.
* eGFR < 30 ml(/min*1.73m2) at baseline.
* Serum potassium > 5.4 mmol/L at baseline.
* Contraindication of ACEI or ARB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Composite outcomes of all-cause death including cardiac death and re-hospitalization due to heart failure

SECONDARY OUTCOMES:
Six-minutes walking test | Test in 1, 3, 6, 12 months comparing to the baseline.
  A test evaluating cardiac function.
LVEF | Test in 1, 3, 6, 12 months comparing to the baseline.
  Left ventricular ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Yihui Xiao, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China